CLINICAL TRIAL: NCT04162314
Title: The Role of β-1,3/1,6-D-Glucan From Extract of Indonesian Ganoderma Lucidum Mycelium as a Combination Therapy With Methylprednisolone for Treatment of Non-infectious and Idiopathic Uveitis: A Double-blind Randomized Pilot Study
Brief Title: Beta-1,3/1,6-D-Glucan Ganoderma Lucidum on Non-infectious and Idiopathic Uveitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Hasianalumban, Ophthalmology resident, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-08-1046
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Uveitis
Keywords: non-infectious uveitis; idiopathic uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): This group received combination of mycelium extract of Ganoderma lucidum capsule containing 180 mg Beta-1,3/1,6-D-Glucan with 3x1 dosage and methylprednisolone (0.8 mg/kgBW) 1x1 for 90 days
  Interventions: Drug: Beta-1,3/1,6-D-Glucan Ganoderma lucidum
- Control (Placebo Comparator): This group received combination of placebo capsules with 3x1 dosage and methylprednisolone (0.8 mg/kgBW) 1x1 for 90 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Beta-1,3/1,6-D-Glucan Ganoderma lucidum — Beta-1,3/1,6-D-Glucan capsule three times daily for 90 days
  Other Names: PsP
  Arms: Experimental
Drug: Placebos — Placebos
  Arms: Control

SUMMARY:
To investigate the effect of Beta-1,3/1,6-D-Glucan from mycelium extract of Indonesian Ganoderma lucidum as an adjuvant to methylprednisolone for non-infectious and idiopathic uveitis

DETAILED DESCRIPTION:
Patients with non-infectious and idiopathic uveitis will receive standard treatment with methylprednisolone, but will be randomized to receive either Beta-1,3/1,6-D-Glucan from mycelium extract of Indonesian Ganoderma lucidum or placebo. Follow up will be performed on week-2, week-4, week-6, month-2, and month-3. Outcomes measured are anterior chamber cells, visual acuity, and serum TNF-alpha levels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-infectious and idiopathic uveitis.
2. Indicated to receive oral steroid and have signs of anterior segment inflammation.
3. Anterior chamber inflammation >= +2 according to SUN criteria.
4. Age between 18 and 65 years old, good general condition, consented to be involved in the research, and are willing to come regularly according to follow up schedule.

Exclusion Criteria:

1. Received systemic steroid and/other immunosuppressive drugs two weeks before the start of the trial.
2. Received antibiotics one week before the start of the trial.
3. Contraindicated to oral steroid.
4. Other primary ocular disorder, such as glaucoma, anterior segment dysgenesis, or others.
5. Pregnant and nursing women.
6. Patients with history of hypersensitivity/ allergy to Ganoderma species or other fungi.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in anterior chamber inflammatory cells grading | Baseline, week-2, week-4, week-6, month-2, month-3
  Change in anterior chamber inflammatory cells grading according to SUN nomenclature (0, 0.5+, 1+, 2+, 3+, 4+). 0 is minimum value (better outcome) and +4 is maximum value (worse outcome).
Change of serum TNF-alpha level | Baseline, week-6, month-3
  Change of serum TNF-alpha level

CONTACTS AND LOCATIONS:
Overall Officials: Lukman Edwar, SpM(K), Dr, Principal Investigator — FKUI/RSCM
Locations (1):
- RSCM Kirana, Jakarta Pusat, DKI Jakarta, Indonesia